CLINICAL TRIAL: NCT00398450
Title: A Phase I Study of 5-azacytidine (Vidaza) With Interferon α2b in Metastatic Melanoma Patients
Brief Title: Azacitidine and Interferon Alfa in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gregory Daniels, Professor, University of California, San Diego
Purpose: Treatment
Other Study IDs: UCSD-060199; CDR0000511743 (Registry Identifier: PDQ (Physician Data Query)); PHARMION-UCSD-060199
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Introns; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: recombinant interferon alfa-2b
Drug: azacitidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Interferon alfa may interfere with the growth of tumor cells. Giving azacitidine together with interferon alfa may be an effective treatment for melanoma.

PURPOSE: This phase I trial is studying the side effects and best dose of azacitidine when given together with interferon alfa in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of azacitidine in combination with interferon alfa-2b in patients with metastatic melanoma.
* Determine if the MTD of this regimen is biologically active in these patients.
* Define and describe the toxicities associated with this regimen.

Secondary

* Determine, preliminarily, the response in patients treated with this regimen.
* Describe, preliminarily, the time to progression and overall survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of azacitidine.

Patients receive azacitidine subcutaneously (SC) once daily on days 1-5 (week 1) followed by interferon alfa-2b SC 3 days a week in weeks 2-4. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of azacitidine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma
* At least one lesion appropriate for 3 separate punch or core needle biopsies
* Must have received and failed ≥ 1 prior systemic treatment for metastatic disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT < 2 times ULN
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known allergies to azacitidine, interferon alfa, benzyl alcohol, or mannitol
* No uncontrolled infection
* No known HIV positivity
* No hepatitis B or hepatitis C infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior systemic therapy
* More than 4 weeks since prior radiotherapy to target lesions with evidence of progression
* No concurrent radiotherapy to target lesions
* No concurrent oral or IV corticosteroids

  * Topical creams or ocular steroid drops are allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Toxicity

SECONDARY OUTCOMES:
Response
Survival at day 1, 12 months, 3 years, and 5 years
Relapse-free survival
Time to relapse

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Daniels, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Rebecca and John Moores UCSD Cancer Center, La Jolla, California, United States